CLINICAL TRIAL: NCT00865553
Title: Clinical Testing of a Decision Support System for Tobacco Use Treatment
Brief Title: Computer-Assisted Stop-Smoking Program in Helping Doctors Counsel Patients Who Smoke Cigarettes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Theodore W. Marcy, Vermont Cancer Center at University of Vermont
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Health Services Research
Other Study IDs: CDR0000629824; VCC-08186; IRB#00000486
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2011-03

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco use disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Early Intervention, Educational

INTERVENTIONS:
Behavioral: computer-assisted smoking cessation intervention
Other: cancer prevention
Other: educational intervention
Other: survey administration

SUMMARY:
RATIONALE: A computer-assisted stop-smoking program may help doctors counsel patients who smoke and may help increase the number of patients who stop smoking.

PURPOSE: This phase II trial is studying how well a computer-assisted stop-smoking program works in helping doctors counsel patients who smoke cigarettes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Test the hypothesis that the clinical decision support system will improve the rate at which physicians assist their patients with smoking cessation by providing information and recommendations on smoking cessation resources.
* Assess whether exposure to information and recommendations facilitated by the smoking cessation-personal digital assistant (SC-PDA) will increase the rate at which patients make at least 1 attempt to quit smoking in the month following the physician visit.
* Assess whether exposure to information and recommendations facilitated by the SC-PDA will increase the reported use of counseling and pharmacotherapy during those attempts over that observed with a smoking status identification system alone.
* Evaluate the acceptance of the SC-PDA into the workflow of ambulatory care clinics.

OUTLINE: In weeks 1-12, physicians have access to a smoking status identification system (SSID) that reminds the physician the smoking status of the patient they are evaluating. In weeks 6-12, physicians have access to a computerized smoking cessation clinical decision support system using a hand-held personal digital assistant (SC-PDA) that they can use in the exam room with their patients who smoke. The SC-PDA system assists physicians in recommending and prescribing approved pharmacotherapy; facilitates referral of patients to local counseling resources; prints a tailored handout for a patient listing specific recommendations, instructions, and cessation resources; and generates the necessary documentation to support billing for this intervention.

Patients who visit their physician in weeks 2-6 or weeks 8-12 complete a survey after their clinic visit and undergo a telephone interview 1 month later. Physicians undergo interviews and focus groups are conducted with clinic staff in weeks 12-16.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Current smoker, defined as self-reported smoking most days or every day (patient)
* Seeks care at a participating Fletcher Allen Health Care primary care clinic (patient)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Physician adherence to the United States Public Health Service's Tobacco Use and Dependence Treatment guideline (USPHS Guideline) as measured by the patient exit survey
Patient perception of physician as measured by the patient exit survey and telephone interview
Prevalence of smoking and associated variables as measured by the patient exit survey
Patient interaction with the smoking cessation-personal digital assistant (SC-PDA) as measured by the patient exit survey and telephone interview
Patient report of physician SC-PDA use as measured by the patient exit survey and telephone interview
Aggregate data on accessing SC-PDA screens by each physician as measured by the SC-PDA server log
Generation of patient handouts as measured by the SC-PDA server log, clinic staff focus groups, and telephone interview
Physician self-reported use of SC-PDA as measured by physician interview
Physician opinion on perceived value and barriers to use as measured by physician interview
Clinic staff opinion on the effect of SC-PDA on clinic workflow as measured by clinic staff focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Theodore W. Marcy, MD, MPH, Principal Investigator — University of Vermont
Locations (1):
- Vermont Cancer Center at University of Vermont, Burlington, Vermont, United States